CLINICAL TRIAL: NCT01866293
Title: A Phase I/II Trial of Cabozantinib (XL184) in Patients With Relapsed or Refractory Myeloma
Brief Title: Cabozantinib (XL184) in Patients With Relapsed or Refractory Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-240
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-02

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Cabozantinib (XL184); 12-240
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — cabozantinib

ARMS (1):
- Cabozantinib (XL184) (Experimental): Eligible patients will receive cabozantinib as a tablet, orally daily. One cycle is defined as 28 days. Myeloma response will be assessed by IMWG criteria after each cycle. The DLT evaluation period will be six weeks. This trial will be a standard 3 by 3 dose escalation design, where three daily dose levels (20mg, 40mg, and 60mg) will be investigated.
  Interventions: Drug: Cabozantinib (XL184)

INTERVENTIONS:
Drug: Cabozantinib (XL184)

SUMMARY:
This study is an open label phase I/II trial to investigate the safety and efficacy of Cabozantinib for patients with relapsed or refractory myeloma.

ELIGIBILITY:
Inclusion Criteria:

* MSKCC confirmed diagnosis of multiple myeloma that has relapsed or is resistant after therapy with at least one immunomodulatory drug (i.e. lenalidomide, thalidomide) and at least one proteasome inhibitor.
* Age ≥ 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

The subject has organ and marrow function as follows:

* Absolute neutrophil count (ANC) ≥ 1500/mm3 (G-CSF is allowed).
* Platelets ≥ 50,000/mm3 or 30,000 (if marrow infiltrated with myeloma; no platelet transfusions are allowed in the 7 days prior to screening)
* Hemoglobin ≥ 8 g/dL (with transfusions). Bilirubin ≤ 1.5 × the upper limit of normal (ULN).
* Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥ 50 mL/min.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN if no liver involvement, or ≤ 5 × ULN with liver involvement.
* Lipase < 1.5 x the upper limit of normal.
* Patient must be able/willing to undergo bone marrow aspirate and biopsy.
* Subjects with brain metastasis or CNS disease are considered eligible if the subject has not received radiation therapy for brain metastasis within 2 weeks of enrollment and has been on a stable dose of steroids for 2 or more weeks.
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g. male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control.
* Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Postmenopause is defined as:
* Amenorrhea ≥ 12 consecutive months without another cause OR
* A documented serum follicle-stimulating hormone (FSH) level > 35 mIU/mL (for women with irregular menstrual periods and on hormone replacement therapy)

Exclusion Criteria:

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 2 weeks, or nitrosoureas/ mitomycin C within 6 weeks before the first dose of study treatment.
* The subject has received radiation therapy within 14 days of the first dose of study treatment.
* The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment.
* The subject has not recovered from toxicity due to all prior therapies (i.e., return to pretherapy baseline or to Grade 0 or 1).
* The subject has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test results at screening that are ≥1.3 ×ULN.
* The subject has uncontrolled significant intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled congestive heart failure, unstable angina pectoris within 6 months, stroke within 6 months, myocardial infarction within 6 months, or uncontrolled cardiac arrhythmias, uncontrolled hypertension.
* Corrected QTc of greater than 500msec.
* The subject is pregnant or breastfeeding.
* The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation.
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel). Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted.
* The subject has experienced any of the following within 6 months before the first dose of study treatment:

  1. clinically-significant hematemesis or gastrointestinal bleeding
  2. hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood
  3. any other signs indicative of pulmonary hemorrhage The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has tumor in contact with, invading or encasing major blood vessels
* Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:
* Any of the following at the time of screening i) intra-abdominal tumor/metastases invading GI mucosa ii) active peptic ulcer disease, iii) inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis iv) malabsorption syndrome

Any of the following within 6 months before the first dose of study treatment:

i) history of abdominal fistula ii) gastrointestinal perforation iii) bowel obstruction or gastric outlet obstruction iv) intra-abdominal abscess. Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 6 months ago.

* History of major surgery as follows:

  1. Major surgery within 3 months of the first dose of cabozantinib. Major surgery within 6 months of the first dose of cabozantinib if there are complications related to wound healing.
  2. Minor surgery within 1 month of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications (particularly when associated with delayed or incomplete healing) within 28 days. Note: Complete healing following abdominal surgery must be confirmed prior to initiating treatment with cabozantinib even if surgery occurred more that 28 days ago.
* Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy or concurrent evidence of intraluminal tumor involving the trachea and esophagus.
* Concurrent malignancy except for treated non-melanoma skin cancer and cervical carcinoma in situ.
* The subject requires chronic concomitant treatment of strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05-28; Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 05/28/2013 Protocol Closed to Accrual 09/16/2015 Primary Completion Date 08/18/2016 Recruitment Location is the medical clinic
Groups:
- Cabozantinib (XL184): Eligible patients will receive cabozantinib as a tablet, orally daily. One cycle is defined as 28 days. Myeloma response will be assessed by IMWG criteria after each cycle. The DLT evaluation period will be six weeks. This trial will be a standard 3 by 3 dose escalation design, where three daily dose levels (20mg, 40mg, and 60mg) will be investigated.
  Cabozantinib (XL184)
Period: Overall Study
Arm/Group | Cabozantinib (XL184)
Started | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 63 [53 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose
Description: This trial will be a standard 3 by 3 dose escalation design, where three daily dose levels (20mg, 40mg, and 60mg) will be investigated.
Time Frame: 1 year
Population: 9 participants are evaluable. 2 participants never started treatment.
Measure: Number; unit: mg
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 11
mg | 40

2. Secondary Outcome: Overall Response Rate
Description: IMWG Criteria for Response, Progression and Relapse in Multiple Myeloma Patients
Time Frame: 1 year
Population: 9 participants are evaluable. 2 participants never started treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 11
Participants
  Progression of disease | 2
  Stable disease | 6
  N/A - off study before disease evaluation | 1
  Did not start study treatment | 2

3. Secondary Outcome: Safety and Toxicity in This Patient Population
Description: Safety assessments and toxicity grading will follow CTCAE Version 4 Grade
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 11
Participants
  Evaluable | 9
  Unevaluable - Enrolled but never started treatment | 2

4. Secondary Outcome: Time to Progression (TTP)
Time Frame: 1 year
Population: 9 participants are evaluable. 2 participants never started treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 11
days | 57 [28 to 85]

5. Secondary Outcome: Duration of Response (DOR)
Time Frame: 1 year
Population: 9 participants are evaluable. 2 participants never started treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 11
days | 63.5 [43 to 85]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cabozantinib (XL184)
All-Cause Mortality (participants affected / at risk) | 5/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (XL184) (N=11)
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 1
Heart failure (Cardiac disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (XL184) (N=11)
Fatigue (General disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Pain (General disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Blood and lymphatic system disorders - Other, spec (Blood and lymphatic system disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysphasia (Nervous system disorders) | 1
Esophageal ulcer (Gastrointestinal disorders) | 1
Gen disorders & admin site conditions Other, spec (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Heart failure (Cardiac disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Irritability (General disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mucosal infection (Infections and infestations) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Urine output decreased (Investigations) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes